CLINICAL TRIAL: NCT03558646
Title: Impact of Hydroxocobalamine on Outcome of Smoke Inhalation Injury Admitted to the ICU
Acronym: COB-AKI
Status: Completed | Type: Observational
Sponsor: Saint-Louis Hospital, Paris, France (Other)
Responsible Party: Principal Investigator, Dr François Dépret, Chef de clinique assistant of the surgical critical burn unit, Principal investigator, Saint-Louis Hospital, Paris, France
Other Study IDs: StLouisFrance01
Record Dates: First submitted 2018-06-01; First posted 2018-06-15 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Smoke Inhalation Patients
Keywords: Smoke inhalation injury; Acute kidney injury; Intensive care unit; Burns; Prognosis; Hydroxocobalamin
MeSH Terms: conditions — Smoke Inhalation Injury; Acute Kidney Injury; Burns

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: There is no intervention planned (observational) — There is no intervention planned (observational)

SUMMARY:
In Europe, hydroxocobalamin (cyanokit) has been used for suspicion of cyanide intoxication associated with the inhalation of fire smoke (1). However, the impact of hydroxocobalamin on outcome has never been thoroughly evaluated. While hydroxocobalamin has long been presented as being side-effect free, recent data suggest that in patients with severe burns, its use was associated with the occurrence of acute renal failure by intra tubular precipitation of oxalate crystals (2, 3). The purpose of this observational study is to investigate the association between use of hydroxocobalamin and outcome after smoke inhalation.

DETAILED DESCRIPTION:
In Europe, hydroxocobalamin (cyanokit) is the antidote recommended by expert consensus in cases of suspicion of cyanide intoxication associated with the inhalation of fire smoke (1). However, cyanokit has never been evaluated in this indication. Clinical data suggest that in patients with severe burns, its use is associated with the occurrence of acute kidney injury by intra tubular precipitation of oxalate crystals (2, 3). The purpose of this observational study is to investigate the association between use of hydroxocobalamin and outcome after smoke inhalation. The results of this study should guide future research and advice on the benefit-risk ratio of hydroxocobalamin.

ELIGIBILITY:
Inclusion Criteria:

* Admission in ICU with smoke inhalation diagnosed

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with smoke inhalation injury admitted in ICU
Sampling Method: Probability Sample
Enrollment: 739 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
in ICU mortality | through study completion, an average of 1 year
  mortality in ICU or at day 90

SECONDARY OUTCOMES:
in ICU acute kidney injury (based on the KDIGO definition) | through study completion, an average of 1 year
  AKI in ICU or at day 90

OTHER OUTCOMES:
Major Adverse Kidney Events | through study completion, an average of 1 year
  MAKE in ICU or at day 90
in ICU length of stay alive | through study completion, an average of 1 year
  through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Saint-Louis Hospital, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. Anseeuw K, Delvau N, Burillo-Putze G, et al.: Cyanide poisoning by fire smoke inhalation: a European expert consensus. Eur J Emerg Med 2013; 20:2-9 2. for the PRONOBURN Study Group, Legrand M, Michel T, et al.: Risk of oxalate nephropathy with the use of cyanide antidote hydroxocobalamin in critically ill burn patients. Intensive Care Medicine 2016; 42:1080-1081 3. Legrand M, Michel T: Empiric use of hydroxocobalamin in patients with smoke inhlation injury: Not so fast! Burns 2017; 43:886
- [Derived] Depret F, Hoffmann C, Daoud L, Thieffry C, Monplaisir L, Creveaux J, Annane D, Parmentier E, Mathieu D, Wiramus S, Demeure DIt Latte D, Kpodji A, Textoris J, Robin F, Klouche K, Pontis E, Schnell G, Barbier F, Constantin JM, Clavier T, du Cheyron D, Terzi N, Sauneuf B, Guerot E, Lafon T, Herbland A, Megarbane B, Leclerc T, Mallet V, Pirracchio R, Legrand M. Association between hydroxocobalamin administration and acute kidney injury after smoke inhalation: a multicenter retrospective study. Crit Care. 2019 Dec 23;23(1):421. doi: 10.1186/s13054-019-2706-0. PMID 31870461